CLINICAL TRIAL: NCT05598008
Title: The Desire PLUS Study - Effects of Glucagon-like-Peptide-1 Analogues on Sexuality: a Prospective Open-label Study
Brief Title: Effects of Glucagon-like-Peptide-1 Analogues on Sexuality
Acronym: Desire PLUS
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-01367; kt22Winzeler
Record Dates: First submitted 2022-10-19; First posted 2022-10-28 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Sexual Desire
Keywords: Glucagon-like-Peptide-1 (GLP-1); Glucagon-like peptide-1 (GLP-1) analogues; obesity; sexuality; Liraglutide (Saxenda®); obese men; reproductive axis; microvascular endothelial function; retinal vessels; physical activity; physical fitness; mood; sperm cells
MeSH Terms: conditions — Obesity; Sexuality; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — If the participant has agreed on further use of biological material blood samples will be stored for an indefinite period of time at - 80°C in a thermo-controlled ultra-deep freezer for eventual future research aims (Biobank department of Endocrinology).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GLP-1 Group: GLP-1 Group: receiving GLP-1 analogues for weight management in addition to conventional weight management (= lifestyle intervention plus GLP-1 analogues).
  Conventional weight management is conducted according to clinical guidelines (in both groups) and includes nutritional and exercise counselling, counselling by motivational coaches and/ or psychological support.
  Participants in the GLP-1 group will inject the medication themselves.
- Lifestyle group: Lifestyle group: using conventional weight management (= lifestyle intervention only).
  Conventional weight management is conducted according to clinical guidelines (in both groups) and includes nutritional and exercise counselling, counselling by motivational coaches and/ or psychological support.

SUMMARY:
This study is to investigate the effects of GLP-1 analogues (combined with lifestyle interventions in comparison to lifestyle interventions only) on sexual desire, mood, quality of life, the reproductive axis, retinal vessel diameters, physical fitness (and semen, for men only) in overweight or obese men and women.

DETAILED DESCRIPTION:
Glucagon-like peptide-1 (GLP-1) analogues are widely used for the treatment of type 2 diabetes mellitus due to its well-known insulinotropic effects as well as for the treatment of obesity due to its satiation-promoting and appetite- suppressant effects. The GLP-1 analogues are approved in patients with obesity (BMI ≥ 30 kg/m2) or who are overweight (BMI ≥ 27 kg/m2) with additional comorbidities, such as prediabetes, diabetes mellitus type 2, arterial hypertension or dyslipidemia. Beside its influence on the reward for palatable food, several studies have shown that GLP-1 analogues modulate the rewarding effects of addictive drugs such as alcohol, nicotine and cocaine. As a further natural reward, sexual desire could be affected by GLP-1 analogues likewise.

This study investigates the influence of GLP-1 analogues on sexuality in a population of overweight and obese participants. A treatment with a GLP-1 analogue combined with lifestyle modifications for weight reduction will be compared to weight reduction with conventional lifestyle modifications only. In the context of the increasing use of GLP-1 analogues, particularly in young people with reproductive desire, laboratory analyzes of the reproductive axis (hormones and sperm cells) will be part of this study to document a possible influence. Mood changes, physical activity and fitness and effects on microvascular endothelial functioning by measuring diameters of retinal vessels will be further investigated.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 27 kg/m2
* Willingness to lose weight by lifestyle changes only or by lifestyle changes plus GLP-1 analogue treatment as agreed in a routine clinical appointment
* Active sex life (sex with partner or masturbation ≥2x/month)
* Eugonadism:

  * Men: morning total testosterone ≥12mmol/l or free testosterone ≥ 0.198 nmol/l if< 50 years old and ≥ 0.163 if > 50 years old
  * Women: no primary or secondary amenorrhea (inclusive menopause) *Secondary amenorrhea is defined as "absence of menses for more than three months in women who previously had regular menstrual cycles or six months in women who had irregular menses".

Exclusion Criteria:

* Diabetes mellitus, HbA1c ≥ 6,5 %
* Previous use of GLP-1 analogues during last 2 months.
* Exogenous testosterone substitution
* Current illicit drug abuse
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of overweight men and women (BMI ≥ 27 kg/m2), which are seen at the obesity clinic of the University Hospital Basel and who wish to lose weight by lifestyle changes and optionally in combination with liraglutide treatment.
Sampling Method: Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2022-11-25 (Actual); Primary Completion 2025-10-24 (Actual); Study Completion 2025-10-24 (Actual)

PRIMARY OUTCOMES:
Change in the German short version of the Sexual Desire Inventory (SDI-2) total score to assess sexual functioning | At baseline (before start of treatment, at V1) and after 4-6 months of treatment (V2)
  The SDI-2 consists of two items addressing frequency of sexual thoughts or activity, rated by a discrete score ranging from 0 to 7 (0 = not at all; 1 = once a month; 2 = once in two weeks; 3 = once a week; 4 = twice a week; 5 = three to four times a week; 6 = once a day; 7 = several times a day), and eight items rating the strengths of different types of sexual desires, rated by a continuous score ranging from 0 to 8 (0 = no desire to 8 = strong desire). The SDI-2 sum score ranges from 0 to 78. A positive score change indicates improvement of sexual desire.

SECONDARY OUTCOMES:
Change in the International Index of Erectile Function (IIEF-5) for men or Female Sexual Function Index (FSFI) for women questionnaire to assess sexual health and erectile function | At baseline (before start of treatment, at V1) and after 4-6 months of treatment (V2)
  The IIEF-5 is a 15-item self-evaluation scale; it provides pre-post treatment clinic evaluations of erectile function, orgasmic function, sexual desire, satisfaction in sexual intercourse and general satisfaction.
  The FSFI is a 19-item self-reporting questionnaire; it measures dimensions such as desire, arousal, lubrication, orgasm, satisfaction, and pain during sexual activity.
Change in the Patient Health Questionnaire (PHQ) -9 questionnaire to assess mood changes | At baseline (before start of treatment, at V1) and after 4-6 months of treatment (V2)
  The PHQ-9 tool may reflect patients' accounts of their experiences of depression and to assess severity of and treatment response. Each of the 9 items can be scored from 0 (not at all) to 3 (nearly every day).
Change in the Patient Health Questionnaire (EQ-5D-5L) questionnaire to assess quality of life | At baseline (before start of treatment, at V1) and after 4-6 months of treatment (V2)
  The EQ-5D descriptive system comprises five dimensions: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression. The five levels in each dimension are worded as (1) 'not /no problems', (2) 'slight problems', (3) 'moderate problems', (4) 'severe problems', and (5) 'unable to' (mobility, self-care, usual activities), 'extreme' (pain/depression), or 'extremely' (anxiety/depression). The second part of the questionnaire comprises a standard vertical 20-cm VAS that is calibrated from 'the worst health you can imagine' (scored 0) at its base to 'the best health you can imagine' (scored 100) at its apex.
Change in retinal vessel diameters to assess microvascular endothelial functioning | At baseline (before start of treatment, at V1) and after 4-6 months of treatment (V2)
  Change in retinal vessel diameters with the Static Retinal Vessel Analyzer (SVA-T, Imedos Systems UG, Jena, Germany). The system consists of a fundus camera (Topcon TRC NW8) and analyzing software (Visualis 3.2, Imedos Systems UG), allowing non-invasive and non-mydriatic assessment of retinal vessel diameters.
Change in Oxytocin Level (IU) (hormone of the reproductive axis) | At baseline (before start of treatment, at V1) and after 4-6 months of treatment (V2)
  Oxytocin Level (hormone of the reproductive axis) will be measured in the blood.
Change in semen concentration | At baseline (before start of treatment, at V1) and after 4-6 months of treatment (V2)
  Change in semen concentration
Change in peak oxygen consumption during spiroergometry to assess physical fitness | At baseline (before start of treatment, at V1) and after 4-6 months of treatment (V2)
  Change in peak oxygen consumption during spiroergometry
Change in maximum heart rate during spiroergometry | At baseline (before start of treatment, at V1) and after 4-6 months of treatment (V2)
  Change in maximum heart rate during spiroergometry
Change in the Freiburg questionnaire for physical activity (FQPA) | At baseline (before start of treatment, at V1) and after 4-6 months of treatment (V2)
  The questionnaire consists of 12 items and allows a calculation of weighted metabolic equivalent tasks (MET) hours per week. The Physical Activity Questionnaire (FPAQ) is used to measure physical activity. Individuals are considered physically active when they achieved metabolic equivalent tasks (MET) minutes of 600 or more per week.
Change in Testosterone level (nmol/l) (hormone of the reproductive axis) | At baseline (before start of treatment, at V1) and after 4-6 months of treatment (V2)
  Testosterone level (hormone of the reproductive axis) will be measured in the blood.
Change in Estradiol level (pmol/l) (hormone of the reproductive axis) | At baseline (before start of treatment, at V1) and after 4-6 months of treatment (V2)
  Estradiol level (hormone of the reproductive axis) will be measured in the blood.
Change in Sex hormone-binding globulin (SHBG) level (nmol/l) (hormone of the reproductive axis) | At baseline (before start of treatment, at V1) and after 4-6 months of treatment (V2)
  Sex hormone-binding globulin (SHBG) level (hormone of the reproductive axis) will be measured in the blood.
Change in Luteinising hormone (LH) level (U/l) (hormone of the reproductive axis) | At baseline (before start of treatment, at V1) and after 4-6 months of treatment (V2)
  Luteinising hormone (LH) level (hormone of the reproductive axis) will be measured in the blood.
Change in Follicle stimulating hormone (LH) level (U/l) (hormone of the reproductive axis) | At baseline (before start of treatment, at V1) and after 4-6 months of treatment (V2)
  Follicle stimulating hormone level (hormone of the reproductive axis) will be measured in the blood.
Change in Prolactin level (yg/l) (hormone of the reproductive axis) | At baseline (before start of treatment, at V1) and after 4-6 months of treatment (V2)
  Prolactin level (hormone of the reproductive axis) will be measured in the blood immediately (10-20 min) after ejaculation.
Change in semen motility | At baseline (before start of treatment, at V1) and after 4-6 months of treatment (V2)
  Change in semen motility
Change in sperm fragmentation index (percentage of sperm with fragmented DNA) | At baseline (before start of treatment, at V1) and after 4-6 months of treatment (V2)
  Change in sperm fragmentation index (percentage of sperm with fragmented DNA)
Change in body weight (kg) | At baseline (before start of treatment, at V1) and after 4-6 months of treatment (V2)
  Body weight is measured during the bioelectrical impedance analysis. The "InBody 720" device is used to perform the analysis.
Change in body fat mass (%) | At baseline (before start of treatment, at V1) and after 4-6 months of treatment (V2)
  Body fat mass is measured during the bioelectrical impedance analysis. The "InBody 720" device is used to perform the analysis.
Change in total body water (l) | At baseline (before start of treatment, at V1) and after 4-6 months of treatment (V2)
  Total body water is measured during the bioelectrical impedance analysis. The "InBody 720" device is used to perform the analysis.
Change in extracellular water (%) | At baseline (before start of treatment, at V1) and after 4-6 months of treatment (V2)
  Extracellular water is measured during the bioelectrical impedance analysis. The "InBody 720" device is used to perform the analysis.
Change in intracellular water (%) | At baseline (before start of treatment, at V1) and after 4-6 months of treatment (V2)
  Intracellular water is measured during the bioelectrical impedance analysis. The "InBody 720" device is used to perform the analysis.
Change in hip/waist ratio | At baseline (before start of treatment, at V1) and after 4-6 months of treatment (V2)
  Hip/waist ratio is measured during the bioelectrical impedance analysis. The "InBody 720" device is used to perform the analysis.
Change in Basal metabolic rate ((kcal/24h) | At baseline (before start of treatment, at V1) and after 4-6 months of treatment (V2)
  Basal metabolic rate is measured during the bioelectrical impedance analysis. The "InBody 720" device is used to perform the analysis.
Change in visceral fat (%) | At baseline (before start of treatment, at V1) and after 4-6 months of treatment (V2)
  Visceral fat is measured during the bioelectrical impedance analysis. The "InBody 720" device is used to perform the analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Winzeler, Dr. med., Principal Investigator — Endocrinology, Diabetes and Metabolism, University Hospital Basel
Locations (1):
- University Hospital Basel, Endocrinology, Diabetes and Metabolism, Basel, Switzerland